CLINICAL TRIAL: NCT01646333
Title: A Randomized Controlled Trial of Neurocognitive and Supportive Therapy Interventions for Individuals With Parkinson's Disease
Brief Title: A Trial of Neurocognitive and Supportive Therapy Interventions for Individuals With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PT107964
Record Dates: First submitted 2012-07-13; First posted 2012-07-20 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Parkinson's Disease; Mild Cognitive Impairment
Keywords: Parkinson Disease; Mild Cognitive Impairment; Cognition; Executive Function; Learning; Memory; Problem Solving
MeSH Terms: conditions — Parkinson Disease; Cognitive Dysfunction | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Supportive Therapy (Active Comparator): The supportive therapy offers patients and support persons the opportunity to discuss and reflect upon both Parkinson's Disease and non-Parkinson's Disease related problems.
  Interventions: Behavioral: Supportive Therapy
- Memory and Problem-Solving Intervention (Experimental): The memory and problem solving training consists of a day calendar manual and note taking system and problem solving techniques. The neurocognitive memory intervention was adapted from a 6-week manualized day calendar and note taking system previously evaluated in an amnestic MCI sample and a brain tumor sample. The problem solving intervention was adapted from an originally 12-week intervention, which was later adapted into a 6-week brain tumor sample.
  Interventions: Behavioral: Memory and Problem-Solving Intervention

INTERVENTIONS:
Behavioral: Memory and Problem-Solving Intervention — 8 weekly 1 hour sessions of memory compensation and problem-solving strategies
  Arms: Memory and Problem-Solving Intervention
Behavioral: Supportive Therapy — 8 weekly 1 hour sessions of non-directive supportive therapy.
  Arms: Supportive Therapy

SUMMARY:
This randomized, controlled trial (RCT) evaluates the benefits of memory and problem solving training compared to supportive therapy in individuals with Parkinson's Disease with Mild Cognitive Impairment (MCI) and their support persons. Participants will be randomly assigned to receive memory and problem solving training or supportive therapy for 2-months. A 6-month follow up evaluation will establish if benefits remain over time. Impact of these therapies on thinking abilities, physical health, and patient and support person ratings of thinking skills, mood and quality of life will be evaluated. The memory and problem solving training is hypothesized to result in greater improvements and/or stability of function on neuropsychological tests of attention, working memory, learning, and memory skills compared to the supportive therapy condition. Both conditions are hypothesized to result in improved mood and quality of life ratings.

Results from this study will determine whether memory and problem solving therapies and supportive therapy are easily used by and beneficial for individuals with Parkinson's Disease and Mild Cognitive Impairment. If positive benefit is observed, information from this study will be used to further optimize these therapies for larger trials designed to evaluate the value of the therapies for individuals with Parkinson's Disease and their support persons.

DETAILED DESCRIPTION:
The memory and problem solving training consists of a day calendar manual and note taking system and problem solving techniques. The supportive therapy offers patients and support persons the opportunity to discuss and reflect upon both Parkinson's Disease and non-Parkinson's Disease related problems.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Parkinson's Disease
* Clinical diagnosis of Mild Cognitive Impairment

Exclusion Criteria:

* Clinical diagnosis of Dementia
* Clinical diagnosis of other Parkinson's Disease-associated comorbid conditions (e.g., severe anxiety, depression, excessive daytime sleepiness, or psychosis) that significantly influence cognitive testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-07; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
California Verbal Learning Test-II Long Delay Free Recall Scaled Score Change Over 10 Weeks | Change from Baseline in California Verbal Learning Test-II Long Delay Free Recall Scaled Score at 10 weeks
  Change in California Verbal Learning Test-II Long Delay Free Recall Scaled Score from Baseline and 10 weeks

SECONDARY OUTCOMES:
Linear Analog Scale Assessment Overall Well Being Raw Score Change Over 10 Weeks | Change from Baseline in Linear Analog Scale Assessment Overall Well Being Raw Score at 10 weeks
  Change in Linear Analog Scale Assessment Overall Well Being Raw Score from Baseline and 10 weeks

OTHER OUTCOMES:
California Verbal Learning Test-II Long Delay Free Recall Scaled Score Change Over 6 Months | Change from Baseline in California Verbal Learning Test-II Long Delay Free Recall Scaled Score at 6 months
  Change in California Verbal Learning Test-II Long Delay Free Recall Scaled Score from Baseline and 6 months
Linear Analog Scale Assessment Overall Well Being Raw Score Change Over 6 Months | Change from Baseline in Linear Analog Scale Assessment Overall Well Being Raw Score at 6 months
  Change in Linear Analog Scale Assessment Overall Well Being Raw Score from Baseline and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sarah K Lageman, Ph.D., Principal Investigator — Virginia Commonwealth University; James P Bennett, Jr., M.D., Ph.D., Study Chair — Virginia Commonwealth University
Locations (1):
- VCU Parkinson's and Movement Disorders Center, Richmond, Virginia, United States